CLINICAL TRIAL: NCT06043440
Title: Randomized Control Trial of Oxygen Therapy in Children and Adolescents With Down Syndrome and Obstructive Sleep Apnea
Brief Title: Down Syndrome Obstructive Sleep Apnea
Acronym: DOSA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital of Philadelphia (Other); Rainbow Babies and Children's Hospital (Other); University of Michigan (Other); Children's Hospital Los Angeles (Other); Children's Hospital of The King's Daughters (Other); Seattle Children's Hospital (Other); University of Southern California (Other)
Responsible Party: Principal Investigator, Susan Redline, Proffesor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023P000062
Record Dates: First submitted 2023-08-17; First posted 2023-09-21 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Down Syndrome; Obstructive Sleep Apnea
MeSH Terms: conditions — Down Syndrome; Sleep Apnea, Obstructive | interventions — Oxygen

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxygen plus supportive care (OXT) (Active Comparator): Nocturnal oxygen therapy plus providing patient with healthy sleep habits materials, healthy diet materials and nasal dilators.
  Interventions: Drug: Oxygen
- Supportive care (SC) (No Intervention): Providing patient with healthy sleep habits materials, healthy diet materials and nasal dilators.

INTERVENTIONS:
Drug: Oxygen — Active nocturnal oxygen concentrator
  Arms: Oxygen plus supportive care (OXT)

SUMMARY:
The purpose of this study is to assess whether oxygen supplementation during sleep improves working memory and other clinical and patient-reported outcomes among children who have Down Syndrome (DS) with moderate to severe Obstructive Sleep Apnea (OSA).

DETAILED DESCRIPTION:
This will be a randomized, single-blind 6-month Phase-2 clinical trial that compares the impact of oxygen therapy during sleep on measures of cognition, behavior, quality of life, cardiac structure and function, and sleep in children with Down Syndrome(DS) with moderate to severe obstructive sleep apnea.

The proposed study will involve participation of children and their caregivers. Children will be recruited from each site's sleep clinics and laboratories, Down syndrome clinics and otolaryngology clinics. Community recruitment will be coordinated with local Down Syndrome Associations.

Children who agree to participate in the study will be screened for eligibility based on history, physical examination, and review of medical records including history of congenital heart disease and Pulmonary Hypertension (PHTN), and use of Continuous Positive Airway Pressure (CPAP). Children eligible for the study are those with persistent obstructive apnea after adenotonsillectomy or children with obstructive sleep apnea without adenotonsillar hypertrophy or in situations when parents refuse adenotonsillectomy.. The enrollment PSG eligibility will be determined by central scoring of either a research Polysomnography (PSG). In addition to an oxygen titration PSG, which determines responsiveness to oxygen, participants will be asked to wear a wrist actigraph and undergo neurocognitive testing, echocardiography, physical examination, anthropometry, and venipuncture. Caregivers will complete questionnaires to assess their child's emotional, physical, social, and school functioning, sleep quality; child's behavior and cognitive function, and will complete a sleep diary that is used concurrently with their child's use of a wrist actigraph. The latter includes caregiver completion of the "Behavior Rating Inventory of Executive Function" (BRIEF2), a co-primary outcome.

At 3 months, caregivers will complete the BRIEF2. At 6 months, all baseline studies and a PSG will be repeated.

At baseline, demographic data will be collected, including information on residential address (for use in geocoding).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 5.0 to 17.9 years at the time of screening
2. Children with OSA and obstructive apnea hypopnea index (OAHI) ≥5/hour.
3. Absence of clinically significant hypoxia defined as oxygen saturation <88% for 5 minutes or episodic desaturation to 60% as these levels would otherwise identify children eligible to routinely receive oxygen.
4. Favorable response to oxygen therapy (allowing randomization) will be defined as follows:

   1. Oxygen saturation nadir >92% and
   2. Decrease in obstructive index < 5 / hour or by > 50% from screening PSG
   3. Reaching an optimum oxygen flow which is defined as the flow that achieves the lowest level of AHI with maximum CO2 level less than 65 mmHg observed for 5 consecutive minutes and or an increase in CO2 by less than 15 points above baseline. The above criteria are observed while the patient spends a minimal of 30 minutes in the supine position and at least one cycle of rapid eye movement (REM) sleep.
   4. Oxygen flow required does not exceed 3.0 LPM and does not exceed a FiO2 > 40 %.
5. Willingness to comply with all study procedures and available for duration of study.
6. At baseline the participant attempts to perform the neuropsychological tests

Exclusion Criteria:

1. Current CPAP use with documented compliance(> 4 hrs/ night; > 70% of nights).
2. Oxygen saturation < 90% at rest during wakefulness.
3. Chronic daytime or nighttime use of supplemental oxygen.
4. Smoker in the child's bedroom.
5. Unrepaired congenital heart disease.
6. Moderate to severe pulmonary hypertension requiring treatment with oxygen and or pulmonary vasodilator.
7. Unable to participate in a PSG.
8. Individuals who develop alveolar hypoventilation with oxygen as previously defined.
9. Other severe chronic diseases determined by their provider as making them poor study candidates.
10. Enrolled or planning to enroll in another study that may conflict with protocol requirements or confound results in this trial.
11. Documented clinically significant untreated hypothyroidism
12. Children with adenotonsillar hypertrophy who are candidates for adenotonsillectomy and parents agree to the surgery.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function 2 (BRIEF2) working memory score | Baseline and 6 months
  Change from baseline in the Behavior Rating Inventory of Executive Function 2 (BRIEF2) working memory score (BRIEF2wm). The score ranges from 35-90. A higher score is a worse outcome.
Differential Ability Scales - 2nd Edition (DAS-II) T-score. | Baseline and 6 months
  Change from baseline in the Differential Ability Scales - 2nd Edition (DAS-II) recognition of pictures (DAS2RoP) T-score. The score ranges from 10-90. A higher score is a better outcome.

SECONDARY OUTCOMES:
Stanford-Binet Intelligence Scales, 5th edition (SB-5) Working Memory Total raw score | Baseline and 6 Months
  Change from baseline of Stanford-Binet Intelligence Scales, 5th edition (SB-5) Working Memory Total raw score. The score ranges from 0-64. A higher score is a better outcome.
Stanford-Binet Intelligence Scales, 5th edition (SB-5) Working Memory Verbal raw score | Baseline and 6 Months
  Change from baseline of Stanford-Binet Intelligence Scales, 5th edition (SB-5) Working Memory Verbal raw score. The score ranges from 0-30. A higher score is a better outcome.
Stanford-Binet Intelligence Scales, 5th edition (SB-5) Working Memory Non Verbal raw score | Baseline and 6 Months
  Change from baseline of Stanford-Binet Intelligence Scales, 5th edition (SB-5) Working Memory Non Verbal raw score. The score ranges from 0-34. A higher score is a better outcome.
Differential Ability Scales-2 (DAS-II) Recall of Digits Forward raw score | Baseline and 6 Months
  Change from baseline in Differential Ability Scales-2 (DAS-II) Recall of Digits Forward raw score. The score ranges from 0-38. A higher score is a better outcome.
Cambridge Neuropsychological Test Automated Battery (CANTAB) Paired Associates Learning (PAL) adjusted total errors based on stages completed | Baseline and 6 Months
  Change from baseline in Cambridge Neuropsychological Test Automated Battery (CANTAB) Paired Associates Learning (PAL) adjusted total errors based on stages completed
Cambridge Neuropsychological Test Automated Battery (CANTAB) Reaction Time (RTI) | Baseline and 6 Months
  Change from baseline in Cambridge Neuropsychological Test Automated Battery (CANTAB) Reaction Time (RTI)
Developmental Neuropsychological Assessment 2nd Edition (NEPSY-II) verbal fluency test raw score | Baseline and 6 Months
  Change from baseline in Developmental Neuropsychological Assessment 2nd Edition (NEPSY-II) verbal fluency test raw score. Range-N/A
Observer Memory Questionnaire - Parent Form (OMQ-PF) total T-score | Baseline and 6 Months
  Change from baseline in Observer Memory Questionnaire - Parent Form (OMQ-PF) total T-score. The score ranges from 0-135. A higher score is a better outcome.
Behavior Rating Inventory of Executive Function 2 (BRIEF2) T-scores for subscales (Inhibit, Self-Monitor, Shift, Emotional Control, Initiate) | Baseline and 6 Months
  Change from baseline in Behavior Rating Inventory of Executive Function 2 (BRIEF2) T-scores for subscales (Inhibit, Self-Monitor, Shift, Emotional Control, Initiate).
Child Behavior Checklist (CBCL) T-scores for domains (Internalizing, Externalizing, Total Problems). | Baseline and 6 Months
  Change from baseline in Child Behavior Checklist (CBCL) T-scores for domains (Internalizing, Externalizing, Total Problems).
Child Behavior Checklist (CBCL) T-scores for subscales (Attention Problems, Thought Problems, Rule-Breaking Behaviors, Aggressive Behaviors) | Baseline and 6 Months
  Change from baseline in Child Behavior Checklist (CBCL) T-scores for subscales (Attention Problems, Thought Problems, Rule-Breaking Behaviors, Aggressive Behaviors)
KIDSCREEN-27 T-score | Baseline and 6 Months
  Change from baseline in KIDSCREEN-27 T-score, including domains of: physical well-being; psychological well-being; autonomy and parent relations; social support and peers; school environment. Range-N/A
Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance T-score | Baseline and 6 Months
  Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance T-score. The score ranges from 28.7-85.6. A higher score is a worse outcome.
Patient-Reported Outcomes Measurement Information System (PROMIS) sleep-related impairment T-score | Baseline and 6 Months
  Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) sleep-related impairment T-score. The score ranges from 37.9-86.6. A higher score is a worse outcome.
Presence of right ventricular hypertension | Baseline and 6 Months
  Presence of right ventricular hypertension as measured by tricuspid regurgitation continuous wave peak velocity (defined as a ratio of pulmonary artery pressure / systolic arterial pressure (PAP/SAP) >1/3); interventricular septal flattening as measured by eccentricity index (defined as systolic ratio of >1.25)
Wechsler Intelligence Scale (WISC) for Children 5th edition (WISC-5) Cancellation raw score | Baseline and 6 Months
  Change from baseline of Wechsler Intelligence Scale (WISC) for Children 5th edition (WISC-5) Cancellation raw score. The score ranges from 0-128. A higher score is a better outcome.
Wechsler Preschool and Primary Scale of Intelligence 4th edition (WPPSI-4) Cancellation task raw score | Baseline and 6 Months
  Change from baseline in Wechsler Preschool and Primary Scale of Intelligence 4th edition (WPPSI-4) Cancellation task raw score (if unable to complete Wechsler Intelligence Scale 5th edition Cancellation test). The score ranges from 0-96. A higher score is a better outcome.
Behavior Rating Inventory of Executive Function 2 (BRIEF2) T-scores for Behavior Regulation Index (BRI) domain. | Baseline and 6 Months
  Change from baseline in Behavior Rating Inventory of Executive Function 2 (BRIEF2) T-scores for Behavior Regulation Index (BRI) domain. The score ranges from 35-90. A higher score is a worse outcome.
Behavior Rating Inventory of Executive Function 2 (BRIEF2) T-scores for Emotional Recognition Index (ERI) domain. | Baseline and 6 Months
  Change from baseline in Behavior Rating Inventory of Executive Function 2 (BRIEF2) T-scores for Emotional Recognition Index (ERI) domain. The score ranges from 35-90. A higher score is a worse outcome.
Behavior Rating Inventory of Executive Function 2 (BRIEF2) T-scores for Cognitive Regulation Index (CRI) domain. | Baseline and 6 Months
  Change from baseline in Behavior Rating Inventory of Executive Function 2 (BRIEF2) T-scores for Cognitive Regulation Index (CRI) domain. The score ranges from 35-90. A higher score is a worse outcome.
7-day actigraphy measurement of sleep efficiency | Baseline and 6 Months
  Change from baseline in 7-day actigraphy measurement of sleep efficiency
7-day actigraphy measurement of time wake after sleep onset | Baseline and 6 Months
  Change from baseline in 7-day actigraphy measurement of time wake after sleep onset
7-day actigraphy measurement of sleep fragmentation | Baseline and 6 Months
  Change from baseline in 7-day actigraphy measurement of sleep fragmentation
7-day actigraphy measurement of total sleep duration | Baseline and 6 Months
  Change from baseline in 7-day actigraphy measurement of total sleep duration
Polysomnography (PSG) AHI parameter | Baseline and 6 Months
  Change from baseline in Polysomnography (PSG) AHI parameter. The score ranges from 0- >40. A higher score is a worse outcome.
Polysomnography (PSG) percentage time of O2 <90 % parameter | Baseline and 6 Months
  Change from baseline in Polysomnography (PSG) percentage time of O2 <90 % parameter
Polysomnography (PSG) sleep apnea associated hypoxic burden parameter | Baseline and 6 Months
  Change from baseline in Polysomnography (PSG) sleep apnea associated hypoxic burden, parameter
Polysomnography (PSG) end-tidal CO2 level, parameter | Baseline and 6 Months
  Change from baseline in Polysomnography (PSG) end-tidal CO2 parameter.
Polysomnography (PSG) -based measure of sleep stages | Baseline and 6 Months
  Change from baseline in Polysomnography (PSG) -based measure of sleep stages. Range- N/A
Polysomnography (PSG) -based measure of EEG power bands | Baseline and 6 Months
  Change from baseline in Polysomnography (PSG) -based measure of EEG power bands
Polysomnography (PSG) -based measure of spindle morphology | Baseline and 6 Months
  Change from baseline in Polysomnography (PSG) -based measure of spindle morphology
Polysomnography (PSG) -based measure of spindle numbers | Baseline and 6 Months
  Change from baseline in Polysomnography (PSG) -based measure of spindle numbers
Polysomnography (PSG) -based measure of spindle density | Baseline and 6 Months
  Change from baseline in Polysomnography (PSG) -based measure of spindle density
Polysomnography (PSG) -based measure of slow wave oscillations | Baseline and 6 Months
  Change from baseline in Polysomnography (PSG) -based measure of slow wave oscillations
Left ventricular diastolic function as measured by Mitral E and A wave (E:A ratio) | Baseline and 6 Months
  Change from baseline in left ventricular diastolic function as measured by Mitral E and A wave (E:A ratio)
Left ventricular diastolic function as measured by E wave deceleration time | Baseline and 6 Months
  Change from baseline in left ventricular diastolic function as measured by E wave deceleration time
Left ventricular diastolic function as measured by Mitral septal and lateral e' and a' (E/e') | Baseline and 6 Months
  Change from baseline in left ventricular diastolic function as measured by Mitral septal and lateral e' and a' (E/e')
Left ventricular diastolic function as measured by Mitral lateral tissue Doppler isovolumic relaxation time | Baseline and 6 Months
  Change from baseline in left ventricular diastolic function as measured by Mitral lateral tissue Doppler isovolumic relaxation time
Left ventricular diastolic function as measured by Pulmonary vein A wave reversal duration | Baseline and 6 Months
  Change from baseline in left ventricular diastolic function as measured by Pulmonary vein A wave reversal duration
Left ventricular diastolic function as measured by Left atrial volume | Baseline and 6 Months
  Change from baseline in left ventricular diastolic function as measured by Left atrial volume

CONTACTS AND LOCATIONS:
Overall Officials: Susan Redline, Principal Investigator — Brigham and Women's Hospital; Raouf Amin, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (7):
- United States (7):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Michigan, Ann Arbor Hospital, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Case Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - East Virginia Medical Center, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Das D, Medina B, Baktir MA, Mojabi FS, Fahimi A, Ponnusamy R, Salehi A. Increased incidence of intermittent hypoxemia in the Ts65Dn mouse model of Down syndrome. Neurosci Lett. 2015 Sep 14;604:91-6. doi: 10.1016/j.neulet.2015.07.040. Epub 2015 Aug 1. PMID 26240993
- [Background] Schloo BL, Vawter GF, Reid LM. Down syndrome: patterns of disturbed lung growth. Hum Pathol. 1991 Sep;22(9):919-23. doi: 10.1016/0046-8177(91)90183-p. PMID 1833304
- [Background] Bush D, Galambos C, Ivy DD, Abman SH, Wolter-Warmerdam K, Hickey F. Clinical Characteristics and Risk Factors for Developing Pulmonary Hypertension in Children with Down Syndrome. J Pediatr. 2018 Nov;202:212-219.e2. doi: 10.1016/j.jpeds.2018.06.031. Epub 2018 Jul 17. PMID 30025669
- [Background] Cooney TP, Wentworth PJ, Thurlbeck WM. Diminished radial count is found only postnatally in Down's syndrome. Pediatr Pulmonol. 1988;5(4):204-9. doi: 10.1002/ppul.1950050405. PMID 2976929
- [Background] Gonzalez OR, Gomez IG, Recalde AL, Landing BH. Postnatal development of the cystic lung lesion of Down syndrome: suggestion that the cause is reduced formation of peripheral air spaces. Pediatr Pathol. 1991 Jul-Aug;11(4):623-33. doi: 10.3109/15513819109064794. PMID 1835001
- [Background] O'Neill AC, Richter GT. Pharyngeal dysphagia in children with Down syndrome. Otolaryngol Head Neck Surg. 2013 Jul;149(1):146-50. doi: 10.1177/0194599813483445. Epub 2013 Mar 22. PMID 23525851
- [Background] Jackson A, Maybee J, Moran MK, Wolter-Warmerdam K, Hickey F. Clinical Characteristics of Dysphagia in Children with Down Syndrome. Dysphagia. 2016 Oct;31(5):663-71. doi: 10.1007/s00455-016-9725-7. Epub 2016 Jul 12. PMID 27405422
- [Background] Khoo MCK, Hu WH, Amin R. Effects of Ventilation-Perfusion Mismatch on Severity of Obstructive Sleep Apnea: A Modeling Study. Annu Int Conf IEEE Eng Med Biol Soc. 2020 Jul;2020:2792-2795. doi: 10.1109/EMBC44109.2020.9175297. PMID 33018586
- [Background] Alex RM, Panza GS, Hakim H, Badr MS, Edwards BA, Sands SA, Mateika JH. Exposure to mild intermittent hypoxia increases loop gain and the arousal threshold in participants with obstructive sleep apnoea. J Physiol. 2019 Jul;597(14):3697-3711. doi: 10.1113/JP277711. Epub 2019 May 9. PMID 31026056
- [Background] Vetrano DL, Carfi A, Brandi V, L'Angiocola PD, Di Tella S, Cipriani MC, Antocicco M, Zuccala G, Palmieri V, Silveri MC, Bernabei R, Onder G. Left ventricle diastolic function and cognitive performance in adults with Down syndrome. Int J Cardiol. 2016 Jan 15;203:816-8. doi: 10.1016/j.ijcard.2015.11.041. Epub 2015 Nov 6. No abstract available. PMID 26595792
- [Background] Mann DM, Esiri MM. The pattern of acquisition of plaques and tangles in the brains of patients under 50 years of age with Down's syndrome. J Neurol Sci. 1989 Feb;89(2-3):169-79. doi: 10.1016/0022-510x(89)90019-1. PMID 2522541
- [Background] Bauer J, Strauss S, Schreiter-Gasser U, Ganter U, Schlegel P, Witt I, Yolk B, Berger M. Interleukin-6 and alpha-2-macroglobulin indicate an acute-phase state in Alzheimer's disease cortices. FEBS Lett. 1991 Jul 8;285(1):111-4. doi: 10.1016/0014-5793(91)80737-n. PMID 1712317
- [Background] Di Domenico F, Tramutola A, Butterfield DA. Role of 4-hydroxy-2-nonenal (HNE) in the pathogenesis of alzheimer disease and other selected age-related neurodegenerative disorders. Free Radic Biol Med. 2017 Oct;111:253-261. doi: 10.1016/j.freeradbiomed.2016.10.490. Epub 2016 Oct 24. PMID 27789292
- [Background] Lyman M, Lloyd DG, Ji X, Vizcaychipi MP, Ma D. Neuroinflammation: the role and consequences. Neurosci Res. 2014 Feb;79:1-12. doi: 10.1016/j.neures.2013.10.004. Epub 2013 Oct 19. PMID 24144733
- [Background] Rueda N, Vidal V, Garcia-Cerro S, Narcis JO, Llorens-Martin M, Corrales A, Lantigua S, Iglesias M, Merino J, Merino R, Martinez-Cue C. Anti-IL17 treatment ameliorates Down syndrome phenotypes in mice. Brain Behav Immun. 2018 Oct;73:235-251. doi: 10.1016/j.bbi.2018.05.008. Epub 2018 May 31. PMID 29758264
- [Background] Rueda Revilla N, Martinez-Cue C. Antioxidants in Down Syndrome: From Preclinical Studies to Clinical Trials. Antioxidants (Basel). 2020 Aug 3;9(8):692. doi: 10.3390/antiox9080692. PMID 32756318
- [Background] Zhang P, Wang Y, Wang H, Cao J. Sesamol alleviates chronic intermittent hypoxia-induced cognitive deficits via inhibiting oxidative stress and inflammation in rats. Neuroreport. 2021 Jan 13;32(2):105-111. doi: 10.1097/WNR.0000000000001564. PMID 33323839
- [Background] Sapin E, Peyron C, Roche F, Gay N, Carcenac C, Savasta M, Levy P, Dematteis M. Chronic Intermittent Hypoxia Induces Chronic Low-Grade Neuroinflammation in the Dorsal Hippocampus of Mice. Sleep. 2015 Oct 1;38(10):1537-46. doi: 10.5665/sleep.5042. PMID 26085297
- [Background] Schmidt-Kastner R. Genomic approach to selective vulnerability of the hippocampus in brain ischemia-hypoxia. Neuroscience. 2015 Nov 19;309:259-79. doi: 10.1016/j.neuroscience.2015.08.034. Epub 2015 Sep 14. PMID 26383255
- [Background] Tietze AL, Blankenburg M, Hechler T, Michel E, Koh M, Schluter B, Zernikow B. Sleep disturbances in children with multiple disabilities. Sleep Med Rev. 2012 Apr;16(2):117-27. doi: 10.1016/j.smrv.2011.03.006. Epub 2011 May 26. PMID 21620745
- [Background] Churchill SS, Kieckhefer GM, Bjornson KF, Herting JR. Relationship between sleep disturbance and functional outcomes in daily life habits of children with Down syndrome. Sleep. 2015 Jan 1;38(1):61-71. doi: 10.5665/sleep.4326. PMID 25325444
- [Background] Edgin JO, Tooley U, Demara B, Nyhuis C, Anand P, Spano G. Sleep Disturbance and Expressive Language Development in Preschool-Age Children With Down Syndrome. Child Dev. 2015 Nov-Dec;86(6):1984-98. doi: 10.1111/cdev.12443. Epub 2015 Oct 5. PMID 26435268
- [Background] Hoffmire CA, Magyar CI, Connolly HV, Fernandez ID, van Wijngaarden E. High prevalence of sleep disorders and associated comorbidities in a community sample of children with Down syndrome. J Clin Sleep Med. 2014 Apr 15;10(4):411-9. doi: 10.5664/jcsm.3618. PMID 24733987
- [Background] Kuroda H, Sawatari H, Ando S, Ohkusa T, Rahmawati A, Ono J, Nishizaka M, Hashiguchi N, Matsuoka F, Chishaki A. A nationwide, cross-sectional survey on unusual sleep postures and sleep-disordered breathing-related symptoms in people with Down syndrome. J Intellect Disabil Res. 2017 Jul;61(7):656-667. doi: 10.1111/jir.12379. Epub 2017 Apr 5. PMID 28378398
- [Background] Pittaras E, Colas D, Chuluun B, Allocca G, Heller C. Enhancing sleep after training improves memory in down syndrome model mice. Sleep. 2022 Apr 11;45(4):zsab247. doi: 10.1093/sleep/zsab247. PMID 34618890
- [Background] Hawkins A, Langton-Hewer S, Henderson J, Tulloh RM. Management of pulmonary hypertension in Down syndrome. Eur J Pediatr. 2011 Jul;170(7):915-21. doi: 10.1007/s00431-010-1378-1. Epub 2011 Jan 4. PMID 21203772
- [Background] Bush D, Abman SH, Galambos C. Prominent Intrapulmonary Bronchopulmonary Anastomoses and Abnormal Lung Development in Infants and Children with Down Syndrome. J Pediatr. 2017 Jan;180:156-162.e1. doi: 10.1016/j.jpeds.2016.08.063. Epub 2016 Sep 22. PMID 27666181
- [Background] Chi TPL?Krovetz J. The pulmonary vascular bed in children with Down syndrome. J Pediatr. 1975 Apr;86(4):533-8. doi: 10.1016/s0022-3476(75)80142-9. PMID 123955
- [Background] Iwaya Y, Muneuchi J, Inoue Y, Watanabe M, Okada S, Ochiai Y. Relationship Between Pulmonary Arterial Resistance and Compliance in Patients with Down Syndrome. Pediatr Cardiol. 2019 Apr;40(4):841-847. doi: 10.1007/s00246-019-02080-9. Epub 2019 Mar 4. PMID 30830280
- [Background] Bush D, Galambos C, Dunbar Ivy D. Pulmonary hypertension in children with Down syndrome. Pediatr Pulmonol. 2021 Mar;56(3):621-629. doi: 10.1002/ppul.24687. Epub 2020 Feb 12. PMID 32049444
- [Background] Amin RS, Kimball TR, Kalra M, Jeffries JL, Carroll JL, Bean JA, Witt SA, Glascock BJ, Daniels SR. Left ventricular function in children with sleep-disordered breathing. Am J Cardiol. 2005 Mar 15;95(6):801-4. doi: 10.1016/j.amjcard.2004.11.044. PMID 15757619
- [Background] Domany KA, Huang G, Hossain MM, Schuler CL, Somers VK, Daniels SR, Amin R. Effect of Adenotonsillectomy on Cardiac Function in Children Age 5-13 Years With Obstructive Sleep Apnea. Am J Cardiol. 2021 Feb 15;141:120-126. doi: 10.1016/j.amjcard.2020.11.019. Epub 2020 Nov 19. PMID 33220319
- [Background] Amin RS, Kimball TR, Bean JA, Jeffries JL, Willging JP, Cotton RT, Witt SA, Glascock BJ, Daniels SR. Left ventricular hypertrophy and abnormal ventricular geometry in children and adolescents with obstructive sleep apnea. Am J Respir Crit Care Med. 2002 May 15;165(10):1395-9. doi: 10.1164/rccm.2105118. PMID 12016102
- [Background] Konstantinopoulou S, Tapia IE, Kim JY, Xanthopoulos MS, Radcliffe J, Cohen MS, Hanna BD, Pipan M, Cielo C, Thomas AJ, Zemel B, Amin R, Bradford R, Traylor J, Shults J, Marcus CL. Relationship between obstructive sleep apnea cardiac complications and sleepiness in children with Down syndrome. Sleep Med. 2016 Jan;17:18-24. doi: 10.1016/j.sleep.2015.09.014. Epub 2015 Oct 23. PMID 26847969
- [Background] Bittles AH, Glasson EJ. Clinical, social, and ethical implications of changing life expectancy in Down syndrome. Dev Med Child Neurol. 2004 Apr;46(4):282-6. doi: 10.1017/s0012162204000441. No abstract available. PMID 15077706
- [Background] Presson AP, Partyka G, Jensen KM, Devine OJ, Rasmussen SA, McCabe LL, McCabe ER. Current estimate of Down Syndrome population prevalence in the United States. J Pediatr. 2013 Oct;163(4):1163-8. doi: 10.1016/j.jpeds.2013.06.013. Epub 2013 Jul 23. PMID 23885965
- [Background] Chamseddin BH, Johnson RF, Mitchell RB. Obstructive Sleep Apnea in Children with Down Syndrome: Demographic, Clinical, and Polysomnographic Features. Otolaryngol Head Neck Surg. 2019 Jan;160(1):150-157. doi: 10.1177/0194599818797308. Epub 2018 Aug 28. PMID 30149781
- [Background] Lee CF, Lee CH, Hsueh WY, Lin MT, Kang KT. Prevalence of Obstructive Sleep Apnea in Children With Down Syndrome: A Meta-Analysis. J Clin Sleep Med. 2018 May 15;14(5):867-875. doi: 10.5664/jcsm.7126. PMID 29734982
- [Background] Cornacchia M, Sethness J, Alapat P, Lin YH, Peacock C. The Prevalence of OSA Among an Adult Population With Down Syndrome Referred to a Medical Clinic. Am J Intellect Dev Disabil. 2019 Jan;124(1):4-10. doi: 10.1352/1944-7558-124.1.4. PMID 30715921
- [Background] Gimenez S, Videla L, Romero S, Benejam B, Clos S, Fernandez S, Martinez M, Carmona-Iragui M, Antonijoan RM, Mayos M, Fortuna A, Penacoba P, Plaza V, Osorio RS, Sharma RA, Bardes I, Rebillat AS, Lleo A, Blesa R, Videla S, Fortea J. Prevalence of Sleep Disorders in Adults With Down Syndrome: A Comparative Study of Self-Reported, Actigraphic, and Polysomnographic Findings. J Clin Sleep Med. 2018 Oct 15;14(10):1725-1733. doi: 10.5664/jcsm.7382. PMID 30353801
- [Background] Gimenez S, Altuna M, Blessing E, Osorio RM, Fortea J. Sleep Disorders in Adults with Down Syndrome. J Clin Med. 2021 Jul 6;10(14):3012. doi: 10.3390/jcm10143012. PMID 34300177
- [Background] Tarasiuk A, Greenberg-Dotan S, Simon-Tuval T, Freidman B, Goldbart AD, Tal A, Reuveni H. Elevated morbidity and health care use in children with obstructive sleep apnea syndrome. Am J Respir Crit Care Med. 2007 Jan 1;175(1):55-61. doi: 10.1164/rccm.200604-577OC. Epub 2006 Oct 12. PMID 17038661
- [Background] Reuveni H, Simon T, Tal A, Elhayany A, Tarasiuk A. Health care services utilization in children with obstructive sleep apnea syndrome. Pediatrics. 2002 Jul;110(1 Pt 1):68-72. doi: 10.1542/peds.110.1.68. PMID 12093948
- [Background] Tarasiuk A, Simon T, Tal A, Reuveni H. Adenotonsillectomy in children with obstructive sleep apnea syndrome reduces health care utilization. Pediatrics. 2004 Feb;113(2):351-6. doi: 10.1542/peds.113.2.351. PMID 14754948
- [Background] Bergeron M, Duggins AL, Cohen AP, Leader BA, Ishman SL. The impact of persistent pediatric obstructive sleep apnea on the Quality of Life of Patients' families. Int J Pediatr Otorhinolaryngol. 2020 Feb;129:109723. doi: 10.1016/j.ijporl.2019.109723. Epub 2019 Oct 12. PMID 31678898
- [Background] Jensen KM, Sevick CJ, Seewald LAS, Halbower AC, Davis MM, McCabe ERB, Kempe A, Abman SH. Greater risk of hospitalization in children with Down syndrome and OSA at higher elevation. Chest. 2015 May;147(5):1344-1351. doi: 10.1378/chest.14-1883. PMID 25654790
- [Background] Boulet SL, Molinari NA, Grosse SD, Honein MA, Correa-Villasenor A. Health care expenditures for infants and young children with Down syndrome in a privately insured population. J Pediatr. 2008 Aug;153(2):241-6. doi: 10.1016/j.jpeds.2008.02.046. Epub 2008 Apr 23. PMID 18534234
- [Background] Kong AM, Hurley D, Evans KA, Brixner D, Csoboth C, Visootsak J. A Retrospective, Longitudinal, Claims-Based Comparison of Concomitant Diagnoses Between Individuals with and Without Down Syndrome. J Manag Care Spec Pharm. 2017 Jul;23(7):761-770. doi: 10.18553/jmcp.2017.23.7.761. PMID 28650250
- [Background] Baker AB, Farhood Z, Brandstetter KA, Teufel RJ 2nd, LaRosa A, White DR. Tonsillectomy in Children with Down Syndrome: A National Cohort of Inpatients. Otolaryngol Head Neck Surg. 2017 Sep;157(3):499-503. doi: 10.1177/0194599817711377. Epub 2017 Aug 1. PMID 28762292
- [Background] Nation J, Brigger M. The Efficacy of Adenotonsillectomy for Obstructive Sleep Apnea in Children with Down Syndrome: A Systematic Review. Otolaryngol Head Neck Surg. 2017 Sep;157(3):401-408. doi: 10.1177/0194599817703921. Epub 2017 May 9. PMID 28485249
- [Background] Propst EJ, Amin R, Talwar N, Zaman M, Zweerink A, Blaser S, Zaarour C, Luginbuehl I, Karsli C, Aziza A, Forrest C, Drake J, Narang I. Midline posterior glossectomy and lingual tonsillectomy in obese and nonobese children with down syndrome: Biomarkers for success. Laryngoscope. 2017 Mar;127(3):757-763. doi: 10.1002/lary.26104. Epub 2016 Jun 27. PMID 27345007
- [Background] Merrell JA, Shott SR. OSAS in Down syndrome: T&A versus T&A plus lateral pharyngoplasty. Int J Pediatr Otorhinolaryngol. 2007 Aug;71(8):1197-203. doi: 10.1016/j.ijporl.2007.04.009. Epub 2007 May 29. PMID 17532478
- [Background] Thottam PJ, Trivedi S, Siegel B, Williams K, Mehta D. Comparative outcomes of severe obstructive sleep apnea in pediatric patients with Trisomy 21. Int J Pediatr Otorhinolaryngol. 2015 Jul;79(7):1013-6. doi: 10.1016/j.ijporl.2015.04.015. Epub 2015 Apr 28. PMID 25959405
- [Background] Europe, K.G., The KIDSCREEN Questionnaires. Quality of life Questionnaires for Children and Adolescents. Lengerich. Pabst Science, 2006.
- [Background] Jennison C and Turnbull GW. 2000. Group Sequential Methods with Applications to Clinical Trials. Boca Raton: Chapman & Hall/CRC.
- [Background] Wittes J, Brittain E. The role of internal pilot studies in increasing the efficiency of clinical trials. Stat Med. 1990 Jan-Feb;9(1-2):65-71; discussion 71-2. doi: 10.1002/sim.4780090113. PMID 2345839
- [Background] Gould LA, and Shih WJ. 1992. Sample Size Re-Estimation Without Unblinding for Normally Distributed Outcomes with Unknown Variance. Communications in Statistics. Theory and Methods 21 (10): 2833-53.
- [Background] Friede T and Miller F. 2012. Blinded Continuous Monitoring of Nuisance Parameters in Clinical Trials. Applied Statistics 61 (4): 601-18.